CLINICAL TRIAL: NCT04529161
Title: Changes in Olfactory and Taste Behavior in Overweight / Obese Subjects Undergoing Fasting Mimicking Diet (FMD)
Brief Title: Olfactory and Taste Changes During Fasting Mimicking Diet (FMD)
Acronym: FMD1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniter Onlus (Other)
Collaborators: University of Rome Tor Vergata (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UniterFMD
Record Dates: First submitted 2020-08-18; First posted 2020-08-27 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Diet, Healthy; Obesity; Olfaction Disorders
MeSH Terms: conditions — Obesity; Olfaction Disorders

STUDY DESIGN:
Intervention Model Description: Patients will follow a 6-months period of FMD followed by a 6-months of routinary eating habits (Group A) or viceversa (Group B)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Diet followed by routine eating
  Interventions: Dietary Supplement: Fasting Mimicking Diet (FMD); Dietary Supplement: Routinary diet habits
- Group B (Experimental): Routine eating followed by diet
  Interventions: Dietary Supplement: Fasting Mimicking Diet (FMD); Dietary Supplement: Routinary diet habits

INTERVENTIONS:
Dietary Supplement: Fasting Mimicking Diet (FMD) — The treatment consists in the self-administration of FMD at home - closely followed by the neuropsychologist by phone and by a properly trained nutritionist in the FMD sector - for 5 days a month for 6 consecutive months.
Dietary Supplement: Routinary diet habits — Subjects will follow their routinary eating habits for 6 consecutive months

SUMMARY:
Literature experiences demonstrated the impact of medically-assisted pulsed fasting on olfactory behavior in both the animal and human models and - conversely - the lack of homogeneous results linked - up to now - to administrations of pulsed fasting which are not widely codified.

Thus, objective of this study protocol is to evaluate the olfactory-gustatory aspects and blood patterns of a group of subjects suffering from obesity / overweight after a 6-month period of Fasting Mimicking Diet (FMD) (Group A) - consisting of a caloric restriction regimen - compared to a group of homogeneous subjects observing their own eating habits (Group B) which - according to a "cross-over" model - will undergo FMD in the following semester during which the subjects belonging to Group A will observe their eating habits.

DETAILED DESCRIPTION:
A group of obese and/or overweighted patients who did not pass screening criteria (BMI andor neuropsychological testing) to undergo surgical procedure aimed at reducing weight (grastrectomy, bypass, other…) will follow a 6-month period of FMD followed by 6-month period of routinary eating behaviour (Group A) or viceversa (Group B).

All the patients will undergo - before and after the administration of FMD or the routinary diet habit - a battery of:

* Olfactory test (sniffin' stick test)
* Taste Test (Taste strips)
* Blood Samples including: IGF-1, IGFBP1/3, VEGF, insulin, adiponectin, c reactive protein, plasma ghrelin, serum glucose, alanine aminotransferase (ALT) and aspartate aminotransferase (AST), total cholesterol, triglycerides (TGs), high density lipoprotein (HDL) cholesterol and low-density lipoprotein (LDL) cholesterol, erythrocyte sedimentation rate (ESR), conjugated and unconjugated bilirubin, uraemia, serum creatinine and leptin.
* anthropometeric measures, including height and body weight, BMI, waist circumference (WC), estimation of fat mass (FM, in % and Kg), skeletal muscle mass (MM, in % and Kg) and grade of visceral fat (VF level)

ELIGIBILITY:
Inclusion Criteria:

* subjects excluded from bariatric surgical treatment for failing to neuropsychological tests or for co-morbidities that would excessively increase the intra-operative and/or
* non-responders to any previous dietary / nutritional treatment
* BMI > 25

Exclusion Criteria:

* Subjects under the age of 18 and over 75 years.
* Subjects already undergoing bariatric surgical treatment
* Women who are pregnant or breastfeeding
* Hormonal therapies and / or chemotherapy in place
* Active mental or psychiatric illness
* Addiction to drugs of abuse or alcohol
* other acute or chronic systemic disorders
* Severe hypertension (systolic blood pressure> 200 mm Hg and / or diastolic blood pressure> 105 mm Hg)
* Visual impairment (for completion of neuropsychological tests)
* Inability to complete home FMD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Sniffing stick test change | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  Quantitative screening of olfactory performance
Taste Strips | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  Quantitative assessment of taste performance

SECONDARY OUTCOMES:
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  serum glucose
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  Serum/plasma growth factors: IGF-1
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  Serum/plasma growth factors: IGFBP1/3
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  Serum/plasma growth factors: insulin
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  Serum/plasma growth factors: VEGF
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  plasma ghrelin.
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  Serum/plasma inflammatory markers: adiponectin
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  Serum/plasma inflammatory markers: c reactive protein
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  alanine aminotransferase
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  aspartate aminotransferase
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  total cholesterol
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  triglycerides
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  high density lipoprotein cholesterol
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  low-density lipoprotein cholesterol
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  erythrocyte sedimentation rate
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  conjugated and unconjugated bilirubin
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  uraemia
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  serum creatinine
Incidence of abnormal laboratory tests results | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  leptin
anthropometric measures | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  height
anthropometric measures | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  weight
anthropometric measures | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  body mass index
anthropometric measures | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  waist circumference
anthropometric measures | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  estimation of fat mass
anthropometric measures | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  estimation of skeletal muscle mass
anthropometric measures | From date of randomization until the date of first documented progression, assessed at the 6th and 12 months
  estimation of grade of visceral fat

CONTACTS AND LOCATIONS:
Overall Officials: Marco Alessandrini, MD, Principal Investigator — University of Rome Tor Vergata
Locations (1):
- University of Rome Tor Vergata - UNITER Onlus, Roma, Rome, Italy

REFERENCES:
- [Background] Cameron JD, Goldfield GS, Doucet E. Fasting for 24 h improves nasal chemosensory performance and food palatability in a related manner. Appetite. 2012 Jun;58(3):978-81. doi: 10.1016/j.appet.2012.02.050. Epub 2012 Mar 2. PMID 22387713
- [Background] Palouzier-Paulignan B, Lacroix MC, Aime P, Baly C, Caillol M, Congar P, Julliard AK, Tucker K, Fadool DA. Olfaction under metabolic influences. Chem Senses. 2012 Nov;37(9):769-97. doi: 10.1093/chemse/bjs059. Epub 2012 Jul 25. PMID 22832483
- [Background] Pager J, Giachetti I, Holley A, Le Magnen J. A selective control of olfactory bulb electrical activity in relation to food deprivation and satiety in rats. Physiol Behav. 1972 Oct;9(4):573-9. doi: 10.1016/0031-9384(72)90014-5. No abstract available. PMID 4670856
- [Background] Tong J, Mannea E, Aime P, Pfluger PT, Yi CX, Castaneda TR, Davis HW, Ren X, Pixley S, Benoit S, Julliard K, Woods SC, Horvath TL, Sleeman MM, D'Alessio D, Obici S, Frank R, Tschop MH. Ghrelin enhances olfactory sensitivity and exploratory sniffing in rodents and humans. J Neurosci. 2011 Apr 13;31(15):5841-6. doi: 10.1523/JNEUROSCI.5680-10.2011. PMID 21490225
- [Background] Tschop M, Weyer C, Tataranni PA, Devanarayan V, Ravussin E, Heiman ML. Circulating ghrelin levels are decreased in human obesity. Diabetes. 2001 Apr;50(4):707-9. doi: 10.2337/diabetes.50.4.707. PMID 11289032
- [Background] English PJ, Ghatei MA, Malik IA, Bloom SR, Wilding JP. Food fails to suppress ghrelin levels in obese humans. J Clin Endocrinol Metab. 2002 Jun;87(6):2984. doi: 10.1210/jcem.87.6.8738. PMID 12050284
- [Background] Meyer-Gerspach AC, Wolnerhanssen B, Beglinger B, Nessenius F, Napitupulu M, Schulte FH, Steinert RE, Beglinger C. Gastric and intestinal satiation in obese and normal weight healthy people. Physiol Behav. 2014 Apr 22;129:265-71. doi: 10.1016/j.physbeh.2014.02.043. Epub 2014 Feb 28. PMID 24582673
- [Background] Stafford LD, Welbeck K. High hunger state increases olfactory sensitivity to neutral but not food odors. Chem Senses. 2011 Jan;36(2):189-98. doi: 10.1093/chemse/bjq114. Epub 2010 Oct 26. PMID 20978137
- [Background] Goldstone AP, Prechtl CG, Scholtz S, Miras AD, Chhina N, Durighel G, Deliran SS, Beckmann C, Ghatei MA, Ashby DR, Waldman AD, Gaylinn BD, Thorner MO, Frost GS, Bloom SR, Bell JD. Ghrelin mimics fasting to enhance human hedonic, orbitofrontal cortex, and hippocampal responses to food. Am J Clin Nutr. 2014 Jun;99(6):1319-30. doi: 10.3945/ajcn.113.075291. Epub 2014 Apr 23. PMID 24760977
- [Background] Wei M, Brandhorst S, Shelehchi M, Mirzaei H, Cheng CW, Budniak J, Groshen S, Mack WJ, Guen E, Di Biase S, Cohen P, Morgan TE, Dorff T, Hong K, Michalsen A, Laviano A, Longo VD. Fasting-mimicking diet and markers/risk factors for aging, diabetes, cancer, and cardiovascular disease. Sci Transl Med. 2017 Feb 15;9(377):eaai8700. doi: 10.1126/scitranslmed.aai8700. PMID 28202779
- [Derived] Micarelli A, Mrakic-Sposta S, Vezzoli A, Malacrida S, Caputo S, Micarelli B, Misici I, Carbini V, Iennaco I, Granito I, Longo VD, Alessandrini M. Chemosensory and cardiometabolic improvements after a fasting-mimicking diet: A randomized cross-over clinical trial. Cell Rep Med. 2025 Feb 18;6(2):101971. doi: 10.1016/j.xcrm.2025.101971. PMID 39970875